CLINICAL TRIAL: NCT06838299
Title: Comparative Study Between Two Different Renal Rehabilitation Protocols on Respiratory and Peripheral Muscles Strength in Hemodialysis Patients
Brief Title: Two Different Renal Rehabilitation Protocols in Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Marwa Atta Ahmed, physiotherapist, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hemodialysis
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Hemodialysis
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): I)inspiratory muscle training:
  Inspiratory muscle training at 60% of maximal inspiratory pressure for 30 minutes/ session, 3 days a week, for 3 months Each patient breathes through a separate mouthpiece. The resistance is adjusted at 60% of maximum inspiratory pressure detected from maximum inspiratory pressure meter and is marked on the training device. A single training session consists of five sets, each contains five inspirations with total of twenty five breaths with one minute of recovery between each set. The resistance was adjusted every week to be 60% of the new maximum inspiratory pressure and if it remained the same, the subject continued to train at the level of the previous week
  Aerobic exercise:
  5-minute warm-up before exercise and a 5-minute cool-down following exercise at intensity (40-65%HR reserve) were carried out each time. In addition, the exercise was performed in the first half of the dialysis session over a 3 months period for 3 sessions per week .
  Interventions: Device: aerobic exercise + inspiratory muscle training
- group B (Active Comparator): Resistance exercise:
  Dynamic closed- and open-chain resistance exercises performed by the patients quadriceps and hamstrings muscles . Patients started at 50% of their initial one-repetition maximum (1-RM) with 5 repetitions for each exercise and later progressed to three sets of 8 repetitions at 70% of their 1-RM according to the patient Borg scale of exertion; training loads were increased when patients could comfortably complete three sets with good form.
  inspiratory muscle training: Inspiratory muscle training at 60% of maximal inspiratory pressure for 30 minutes/ session, 3 days a week, for 3 months Each patient breathes through a separate mouthpiece. The resistance is adjusted at 60% of maximum inspiratory pressure detected from maximum inspiratory pressure meter and is marked on the training device. A single training session consists of five sets, each contains five inspirations with total of twenty five breaths with one minute of recovery between each set.
  Interventions: Device: resistance exercise + inspiratory muscle training
- group C (control group) (Active Comparator): in this group there is no exercise ,patients have assessment pre and post 3 months and follow up
  Interventions: Other: control group

INTERVENTIONS:
Device: aerobic exercise + inspiratory muscle training — inspiratory muscle training: Inspiratory muscle training at 60% of maximal inspiratory pressure for 30 minutes/ session, 3 days a week, for 3 months Each patient breathes through a separate mouthpiece. The resistance is adjusted at 60% of maximum inspiratory pressure detected from maximum inspiratory pressure meter and is marked on the training device. A single training session consists of five sets, each contains five inspirations with total of twenty five breaths with one minute of recovery between each set. The resistance was adjusted every week to be 60% of the new maximum inspiratory pressure and if it remained the same, the subject continued to train at the level of the previous week Aerobic exercise: by bicycle ergomete 5-minute warm-up before exercise and a 5-minute cool-down following exercise at intensity (40-65%HR max) were carried out each time. In addition, the exercise was performed in the first half of the dialysis session over a 3 months period for 3 sessions a week
  Arms: group A
Device: resistance exercise + inspiratory muscle training — Resistance exercise:
  Dynamic closed- and open-chain resistance exercises performed by the patients quadriceps and hamstrings muscles . Patients started at 50% of their initial one-repetition maximum (1-RM) with 5 repetitions for each exercise and later progressed to three sets of 8 repetitions at 70% of their 1-RM according to the patient Borg scale of exertion; training loads were increased when patients could comfortably complete three sets with good form.
  inspiratory muscle training: Inspiratory muscle training at 60% of maximal inspiratory pressure for 30 minutes/ session, 3 days a week, for 3 months Each patient breathes through a separate mouthpiece. The resistance is adjusted at 60% of maximum inspiratory pressure detected from maximum inspiratory pressure meter and is marked on the training device. A single training session consists of five sets, each contains five inspirations with total of twenty five breaths with one minute of recovery between each set.
  Arms: group B
Other: control group — there is no exercise , patients do assessment pre and post 3 months and follow up
  Arms: group C (control group)

SUMMARY:
the goal of this clinical trial is to find out the effect of combined inspiratory muscle training with aerobic exercise or combined inspiratory muscle training with resistance exercise for hemodialysis CKD patients .the main question it aims to answer is is There a significant difference in the effect of aerobic exercise or resistance exercise (Inspiratory muscle training and peripheral resistance training) for hemodialysis CKD patients.

researchers will compare effect of (aerobic exercise +inspiratory muscle training),or (resistance exercise +inspiratory muscle training) and control group participants will be at regular hemodialysis of both sex aged from forty to sexty years will be recruited in this study from kidney dialysis department and do exercie 3 times a week for 3 months

DETAILED DESCRIPTION:
Type of study: Randomized controlled trial

This study is a prospective interventional study one that will be conducted on ninty chronic kidney disease patients at regular hemodialysis of both sex aged from forty to sexty years will be recruited in this study from kidney dialysis department and will randomly divided into three equal groups:

1. intervention group 1:include 30 CKD patients at hemodialysis will receive aerobic exercise ,inspiratory muscle training and medical treatment
2. Intervention group 2: include 30 CKD patients at hemodialysis will receive resistance exercise, inspiratory muscle training and medical treatment
3. control group: include 30 CKD patients at hemodialysis will receive medical treatment only

Instrumentations:

• Evaluation will be done before and after treatment and follow up after 3months and 6months from the beginning of treatment.

A)Evaluation equipment

1. Maximum inspiratory pressure meter: (care fusion UK 2321td).
2. Kidney Disease and Quality of Life (KDQOL-SF™ 1.3)
3. Peak oxygen consumption (predicted Peak VO2):

4-6minute walk test. 5-Modified Borg scale (asses The sensation of dyspnea, fatigue of lower limbs during walk) 6- Echo cardiogram to detect left ventricular ejection fraction.

B) training equipment:

1. inspiratory muscle trainer:(Threshold® Inspiratory Muscle Trainer , Calibrated, Spring-Loaded Valve with adjustable pressure from 7 to 41 cm H2O.
2. Bicycle ergometer
3. weight(sand bags)

Evaluation procedures:

1. Maximum inspiratory pressure meter: to determine the inspiratory muscle strength before and after training.

   the patient will be instructed to insert the mouthpiece into the mouth, ensuring the flange is positioned over the gums and inside the lips, while the 'bite blocks' are between the teeth. The subject should then exhale to RV (Residual Volume), then perform a forced inhalation against the mouthpiece with as much effort as possible for as long as possible (minimum 2 seconds). while the participants were seated in a reclining chair (with knees and hips at 90) in a HD room at the beginning of the HD session ( Laveneziana et al,2019)
2. Kidney Disease and Quality of Life (KDQOL-SF™ 1.3): KDQOL-36 is a short version of KDQOL-SFthat includes only 36 questions.2 The survey can be administered in 3-5 min, which saves both time and resources in large-scale population surveys. Each subscale score ranges between 0 and 100, with increasing values equating to better health. (Saudi, 2019)
3. peak vo2: predicted peak vo2 with cahalin equation: Peak vo2 =0.03× distance in meter +3.98, by detecting the walking distance from 6MWT.(Morisheta et al,2017) 4-6-minute walk test : (To detect functional capacity, carry out in a 30-meter line along The passage way, The tape is placed every 2meters.patients are instructed to walk The longest possible distance in 6minutes continuously, turning around at The final Mark without stopping. they are further instructed to walk as far as they can for 6minutes without running or jogging, covered distance in meters is measured at the end of the rest for analysis (Jamshidpour et al,2020)

5-modified Borg scale: asses The sensation of dyspnea, fatigue during exercise (Watanabe et al,2021) 6-one- repetition maximum (1RM) 7-lab analysis) GFR, Serum cretinine, blood urea ) Treatment Procedures Training for 3 months,3sessins per week intradialysis at the first two hours. intervention: I)inspiratory muscle training: for group A and B Inspiratory muscle training at 60% of maximal inspiratory pressure for 30 minutes/ session, 3 days a week, for 3 months Each patient breathes through a separate mouthpiece. The resistance is adjusted at 60% of maximum inspiratory pressure detected from maximum inspiratory pressure meter and is marked on the training device. A single training session consists of five sets, each contains five inspirations with total of twenty five breaths with one minute of recovery between each set. The resistance was adjusted every week to be 60% of the new maximum inspiratory pressure and if it remained the same, the subject continued to train at the level of the previous week (Yuenyongchaiwat et al,2021) 2) Aerobic exercise: for group A 5-minute warm-up before exercise and a 5-minute cool-down following exercise at intensity (30-40%HR max) were carried out each time. In addition, the exercise was performed in the first half of the dialysis session over a 3 months period for 3 sessions per week by cycling for 20 min at a moderate intensity(70-80%HRmax) participants were trained to use stationary bicycle ergometer (Thera-fit Plus bed trainer, Medica Medizintechnik, Hochdorf, Germany) in a supine position for minimum of 30 minutes at each HD session. The speed, load, and duration were gradually increased with change of mode (automatic and passive) and application of sand bags. According to patients' performance, training loads were adjusted (Rhee et al,2019) 3)Resistance exercise: for group B Dynamic closed- and open-chain resistance exercises performed by the patients quadriceps and hamstrings muscles . Patients started at 50% of their initial one-repetition maximum (1-RM) with 5 repetitions for each exercise and later progressed to three sets of 8 repetitions at 70% of their 1-RM according to the patient Borg scale of exertion; training loads were increased when patients could comfortably complete three sets with good form. The training resistance was adjusted according to the newly achieved one-repetition maximum (1-RM)

Purpose of the study:

To find out the effect of combined inspiratory muscle training with aerobic exercise or combined inspiratory muscle training with resistance exercise for hemodialysis CKD patients as regards The following outcomes:

1. medical state of patient (heart rate, blood pressure, oxygen saturation)
2. lab analysis (GFR, Serum cretinine, blood urea and nitrogen (BUN))
3. Inspiratory muscle pressure(MIP,MEP)
4. period, duration of dialysis
5. weight, height, BMI
6. quality of Life questionnaire
7. modified Borg scale

ELIGIBILITY:
Inclusion Criteria:

* Patients from both gender
* With chronic kidney disease
* Unemployed living a sedentary lifestyle
* Receive regular hemodialysis sessions at 3months ago
* All of them have vascular access through arteriovenous fistula
* Age range from 40-60years
* Fully understand purpose and procedure of study
* Stable and have sufficient level of cognition and ability to understand instructions

Exclusion Criteria:

* • Real difficulties with understanding and signing The written informed consent

  * Recent sequela of cerebrovascular accidents
  * Osteoarticular or musculoskeletal diseases
  * Un controlled systemic hypertension
  * Un controlled diabetes
  * Un stable angina
  * Fever
  * Infectious disease
  * Acute respiratory failure
  * Recent acute myocardial infarction
  * Smoking
  * Peripheral vascular alterations

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-05-28 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
6minute walk test | at the start of study , after intervention (after 3 months), and follow up (after 3 months of intervention)
  -6 minute walk test : to detect functional capacity , carry out in a 30 meters line along the passage way , the tape is placed every 2 meter . patients are instructed to walk the longest possible distance in 6 minutes continuously and turning around at the final mark without stopping .they are instructed to walk as far as they can for 6 minutes without running or jogging .covered distance in meters is measured at the end of analysis.

SECONDARY OUTCOMES:
Maximum inspiratory pressure | at the start of study , after intervention (after 3 months), and follow up (after 3 months of intervention)
  -Maximum inspiratory pressure : to determine the inspiratory muscle strength before and after training. the patient will be instructed to insert the mouthpiece into the mouth, ensuring the flange is positioned over the gums and inside the lips, while the 'bite blocks' are between the teeth. The subject should then exhale to RV (Residual Volume), then perform a forced inhalation against the mouthpiece with as much effort as possible for as long as possible (minimum 2 seconds). while the participants were seated in a reclining chair (with knees and hips at 90) in a HD room at the beginning of the HD session .

CONTACTS AND LOCATIONS:
Overall Officials: Sherine H Mehani, professor, Principal Investigator — Beni-Suef University
Locations (1):
- Beni_suef university, Beni_suef, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rhee et al,2019